CLINICAL TRIAL: NCT00149656
Title: HIV Disease, Drug Abuse, and Nutrient Therapy in Botswana
Brief Title: The Effects of Nutritional Supplementation and Drug Abuse on HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-16551-1; R01DA016551 (NIH); R01-16551-1; DPMC
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: HIV Infections; Substance-Related Disorders
Keywords: Treatment Naive; Multivitamins; Selenium; Supplementation; HIV Disease Progression
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders | interventions — Geritol; Selenium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Other: Placebo
- 2 (Experimental): Multivitamins
  Interventions: Dietary Supplement: Multivitamins
- 3 (Experimental): Multivitamins with Selenium
  Interventions: Dietary Supplement: Multivitamins; Dietary Supplement: Selenium
- 4 (Experimental): Selenium
  Interventions: Dietary Supplement: Selenium

INTERVENTIONS:
Dietary Supplement: Multivitamins — dietary supplement of multivitamins
  Arms: 2; 3
Dietary Supplement: Selenium — dietary supplement of selenium only
  Arms: 3; 4
Other: Placebo — placebo pill
  Arms: 1

SUMMARY:
The purpose of this trial is to determine whether supplementation with multivitamins and selenium will delay disease progression in HIV infected individuals in Botswana. The study will also assess how drug abuse modifies the effect of nutritional supplementation on HIV disease progression.

DETAILED DESCRIPTION:
Botswana has the highest rates of HIV infection in the world. In addition, drug abuse has become an emerging problem in Botswana. Past research suggests that multivitamin and selenium supplementation slows the progression of HIV disease. The purpose of this trial is to evaluate the effectiveness of supplementation with multivitamins and selenium in HIV infected individuals in Botswana.

This trial will last 2 years. Participants will be randomly assigned to 4 groups: a combination of multivitamins with selenium, multivitamins alone, selenium alone, or placebo.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* CD4 count greater than 350 cells/mm3
* Identified from the Infectious Disease Care Clinic
* Body mass index greater than 18 for women and greater than 18.5 for men

Exclusion Criteria:

* Current AIDS-defining condition
* Currently participating in another clinical trial
* Pregnant or intends to become pregnant during the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 878 (Actual)
Dates: Start 2003-06; Primary Completion 2010-07 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
HIV Disease Progression | For at least 6 months

SECONDARY OUTCOMES:
Morbidity | For at least 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marianna K. Baum, PhD, Principal Investigator — Florida International University
Locations (1):
- Princess Marina Hospital, Gaborone, Botswana